CLINICAL TRIAL: NCT06338917
Title: Moderate-to-Vigorous Intensity Physical Activity as a Tool for Severe Mental Illness Recuperation Process: Study Protocol for a Pragmatic Controlled Clinical Trial (+moviMENT)
Brief Title: Moderate-to-Vigorous Intensity Physical Activity and Severe Mental Illness
Acronym: +MoviMENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: IRIS-CC (Unknown); AGAUR (Unknown)
Responsible Party: Principal Investigator, Mariona Caro Crous, MsC in physical activity and health and graduate in physical activity and sport science, University of Vic - Central University of Catalonia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: File 2022 DI 61
Record Dates: First submitted 2024-03-13; First posted 2024-04-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue
Keywords: mental illness; exercise; sedentary behaviour; lifestyle
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a pragmatic controlled clinical trial with intervention and control group, in which patients will be recruited from two different services from different cities.
Who Masked: Participant, Care Provider
Masking Description: Participants in both groups are not aware of the existence of the other group. The health provider in the control group is aware of the existence of the intervention group but does not know which intervention is being carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participation in a moderate-to-vigorous intensity physical activity program a part from the usual health care treatment
  Interventions: Behavioral: Moderate-to-vigorous intensity physical activity program (+moviMENT)
- Control group (No Intervention): Following the usual health care treatment

INTERVENTIONS:
Behavioral: Moderate-to-vigorous intensity physical activity program (+moviMENT) — The intervention comprises 16 weeks of group based High Intensity Interval Training (HIIT), with transition to individual community based Vigorous Intermittent Lifestyle Physical Activity (VILPA) over the next 12 weeks - for a total intervention period of 28 weeks.
  Arms: Intervention group

SUMMARY:
Twenty-five percent of the population worldwide will experience a severe mental illness during their lifetime (World Health Organization, 2017). These people present strong barriers to adhering to moderate and vigorous-intensity continuous training. It is fundamental to overcome these barriers for practicing moderate-to-vigorous physical activity by adding behavioural change techniques into physical activity interventions (Maurus et al., 2023), in order to design and implement sustainable interventions that empower people to engage in it.

The overall aims will be to evaluate the efficacy of +moviMENT, a 28-week intervention program, designed to increase MVPA time in patients with SMI, and to assess the effects of the program on a range of indicators, in comparison with a 'usual care' control group.

DETAILED DESCRIPTION:
This is a pragmatic controlled clinical trial with intervention and control group, in which patients will be recruited from two different services from different cities. Patients who will meet the inclusion criteria (>16 years, severe mental illness diagnosis, not medical risk to practice MVPA, living in the community) from one service will be assigned to the intervention and those from the other to the control group. The intervention comprises 16 weeks of group based High Intensity Interval Training (HIIT), with transition to individual community based Vigorous Intermittent Lifestyle Physical Activity (VILPA) over the next 12 weeks - for a total intervention period of 28 weeks. Primary outcomes measures (clinical and functional) and secondary (personal recovery, self-perception and device-measured fitness, physical activity and sedentary behaviour and experience) will be assessed at baseline and after 16, 28 and 40 weeks, after follow-up. Group differences in change scores will be assessed using linear mixed-effects models with time, group, and their interaction as fixed effects, accounting for within-subject correlations.

ELIGIBILITY:
* Outpatients (non-hospitalised) registered in one of two mental health services.
* SMI diagnosis, according to the 5th edition of the 5th Diagnostic and Statistical Manual of mental disorders (DSM-5) [52].
* Living in the community
* Not having any contraindications or medical risk to MVPA.
* Age 18 to 69 years.
* Willing and able to provide informed consent.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Disability | Measurement will be at the beginning, 4, 7 and 10 follow-up months.
  World Health Organization-Disability Assessment Schedule II (WHODAS 2.0): Scale that assesses the activity limitations and participation restrictions experienced by the person. Through its 36 items, the WHODAS II allows us to obtain, both at a specific and general level, a measure of the severity and duration of the disability that results from the "health conditions" of people, also providing information on the "costs" that they generate in the individual, in the family or in society.
Cognitive functioning | Measurement will be at the beginning, 4 and 7 months.
  Screen for Cognitive Impairment in Psychiatry (SCIP-S): This scale is designed to assess cognitive deficits in psychiatric patients. It consists of 5 subtests that assess immediate and delayed verbal learning, working memory, verbal fluency and processing speed. The total score is the sum of the 5 subscales and its interpretation allows detecting the presence of cognitive deficit; a higher score corresponds to better cognitive performance.
Psychotic symptomatology | Measurement will be at the beginning, 4 and 7 months.
  The Brief Psychiatric Rating Scale (BPRS) is a rating scale which a clinician or researcher may use to measure psychiatric symptoms such as depression, anxiety, hallucinations, psychosis and unusual behaviour. It has 18 items. The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe). It is scored by adding together the scores from the individual items, with higher scores indicating more severe symptoms.
Depression symptomatology | Measurement will be at the beginning, 4 and 7 months.
  Hamilton Depression Rating Scale (HAM-D): A 17-item mood rating scale. A score below 7 is considered to indicate no depressed mood, a score between 8 and 16 is considered to be moderate depression and a score above 18 indicates severe depression.

SECONDARY OUTCOMES:
Device-measured physical activity and sedentary behaviour pattern | Measurement will be at the beginning, 4 and 7 months.
  To measure physical activity and sedentary behavior, the activPAL3TM will be used. This is a miniature electronic logger designed to quantify daily free-living activities. With the activPAL3TM you can obtain a record of total sitting time, number of sitting time interruptions, sedentary bouts, standing time and activity time (light, moderate and vigorous-intensity).
Fitness self-perception | Measurement will be at the beginning, 4, 7 and 10 follow-up months.
  The International Fitness Scale (IFIS) evaluates people's perception of physical fitness. It is a 5-item scale (general fitness, cardio-respiratory, muscular strength, speed and agility, and flexibility) rated from 1 to 5, with 1 being "very bad" and 5 being "very good". The final result is obtained from the sum total of the items, with the highest score being 25. The higher the final result, the better the perception.
Quality of life self-perception | Measurement will be at the beginning, 4, 7 and 10 follow-up months.
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health with regard to the respective domain. Thus, the patient's physical, psychological, social, and environmental state of health are assessed separately.
Physical activity pattern self-perception | Measurement will be at the beginning, 4, 7 and 10 follow-up months.
  International Physical Activity Questionnaire, short and Spanish version, (IPAQ-SF17). A 7-question scale that assesses habitual physical activity (minutes/week) performed in the last 7 days. It measures physical activity performed at different intensities: vigorous, moderate and light physical activity. The total physical activity (minutes/week) is obtained from the sum total of the minutes/week of physical activity performed at the different intensities.
Sedentary behaviour pattern self-perception | Measurement will be at the beginning, 4, 7 and 10 follow-up months.
  Sedentary Behavior Questionnaire, Spanish version (SBQ). Scale of 22 items, divided into two blocks: weekdays and weekends. The scale identifies the hours/day spent sitting, stretching or reclining during the day before doing the following activities: watching TV, playing PC/video games, eating, resting while lying down, sitting in a vehicle, doing office work, relaxing (e.g. reading or listening to music). The total daily hours of sedentary behaviour are obtained by adding the hours/day spent in each of the above activities. Total daily hours are obtained for both weekdays and weekends.
Cardiorespiratory endurance | Measurement will be at the beginning, 4 and 7 months.
  The 6-minute walk test is a test in which the person walks at his or her normal pace for 6 minutes. Every minute the person is asked how fatigued he/she is (with the Borg Fatigue Scale). The more meters the person walks, the better the cardio-respiratory condition.
Agility | Measurement will be at the beginning, 4 and 7 months.
  The T-test is a test in which the person has to do a T-shaped circuit as fast as possible, combining forward, backward and sideways movements. When evaluating the test, the speed of execution is taken into account, as well as the correct execution of the movements.
Lower limb strength | Measurement will be at the beginning, 4 and 7 months.
  The sit-to-stand test is a test in which the person has to stand up and sit down on a chair 5 times in a row as fast as possible. The faster the person is able to do the repetitions, the better the evaluation of the test.

OTHER OUTCOMES:
Patient Reported Experience Measures (PREM) and Patient Reported Outcome Measures (PROM) | Measurement will be at the final of the intervention, month 7.
  PREMs (Patient Reported Experience Measures) refer to measures that assess the patient's experience of the care received. These measures are obtained directly from patients through surveys or questionnaires and are used to assess aspects such as communication with health care providers, participation in decision-making, access to health care services, overall satisfaction and other aspects of the patient experience. PROMs (Patient Reported Outcome Measures) focus on the measurement of self-reported outcomes related to their health, symptoms and quality of life. These measures are also obtained directly from patients through surveys or questionnaires and assess aspects such as pain intensity, physical functioning, emotional well-being, sleep quality and other health domains that are relevant to the patient. PROMs provide insight into the patient's perspective on the impact of a disease, treatment or intervention on their daily life and general well-being.
Mood | Measurement will be at the beginning and during all the physical activity sessions.
  Visual analogue subjective mood scale (VAS). A visual scale designed to determine subjective mood state, which can be rated from 0 to 10, with 0 being "I feel worse than ever" and 10 being "I feel better than ever".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vic, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and supplementary material) will be shared. Only IPD used in the results will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available following the publication of the results from the study protocol. No end date.
Access Criteria: Everyone who will be interested in the results of the pragmatic clinical trial will be able to access the IPD. The information shared will be the analysis data set, tables and figures. Readers will be able to access the IPD through supplementary material.

REFERENCES:
- [Background] Chen MD, I JH, Pellegrini CA, Chen HF, Su CY, Chang YC. The facilitators and barriers to physical activity scale for people with mental illness in Taiwan: development and validation. Disabil Rehabil. 2022 Aug;44(17):4879-4887. doi: 10.1080/09638288.2021.1916627. Epub 2021 Apr 25. PMID 33896304
- [Background] Glover CM, Ferron JC, Whitley R. Barriers to exercise among people with severe mental illnesses. Psychiatr Rehabil J. 2013 Mar;36(1):45-7. doi: 10.1037/h0094747. PMID 23477650
- [Background] Thogersen-Ntoumani C, Kritz M, Grunseit A, Chau J, Ahmadi M, Holtermann A, Koster A, Tudor-Locke C, Johnson N, Sherrington C, Paudel S, Maher C, Stamatakis E. Barriers and enablers of vigorous intermittent lifestyle physical activity (VILPA) in physically inactive adults: a focus group study. Int J Behav Nutr Phys Act. 2023 Jul 4;20(1):78. doi: 10.1186/s12966-023-01480-8. PMID 37403160
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Schuch FB, Vancampfort D, Firth J, Rosenbaum S, Ward PB, Silva ES, Hallgren M, Ponce De Leon A, Dunn AL, Deslandes AC, Fleck MP, Carvalho AF, Stubbs B. Physical Activity and Incident Depression: A Meta-Analysis of Prospective Cohort Studies. Am J Psychiatry. 2018 Jul 1;175(7):631-648. doi: 10.1176/appi.ajp.2018.17111194. Epub 2018 Apr 25. PMID 29690792
- [Background] Malchow B, Reich-Erkelenz D, Oertel-Knochel V, Keller K, Hasan A, Schmitt A, Scheewe TW, Cahn W, Kahn RS, Falkai P. The effects of physical exercise in schizophrenia and affective disorders. Eur Arch Psychiatry Clin Neurosci. 2013 Sep;263(6):451-67. doi: 10.1007/s00406-013-0423-2. Epub 2013 Jul 20. PMID 23873090
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] Scheewe TW, Backx FJ, Takken T, Jorg F, van Strater AC, Kroes AG, Kahn RS, Cahn W. Exercise therapy improves mental and physical health in schizophrenia: a randomised controlled trial. Acta Psychiatr Scand. 2013 Jun;127(6):464-73. doi: 10.1111/acps.12029. Epub 2012 Oct 26. PMID 23106093
- [Background] Scheewe TW, Takken T, Kahn RS, Cahn W, Backx FJ. Effects of exercise therapy on cardiorespiratory fitness in patients with schizophrenia. Med Sci Sports Exerc. 2012 Oct;44(10):1834-42. doi: 10.1249/MSS.0b013e318258e120. PMID 22525773
- [Background] Heissel A, Heinen D, Brokmeier LL, Skarabis N, Kangas M, Vancampfort D, Stubbs B, Firth J, Ward PB, Rosenbaum S, Hallgren M, Schuch F. Exercise as medicine for depressive symptoms? A systematic review and meta-analysis with meta-regression. Br J Sports Med. 2023 Aug;57(16):1049-1057. doi: 10.1136/bjsports-2022-106282. Epub 2023 Feb 1. PMID 36731907
- [Background] Garcia-Garces L, Sanchez-Lopez MI, Cano SL, Melia YC, Marques-Azcona D, Bivia-Roig G, Lison JF, Peyro-Gregori L. The short and long-term effects of aerobic, strength, or mixed exercise programs on schizophrenia symptomatology. Sci Rep. 2021 Dec 21;11(1):24300. doi: 10.1038/s41598-021-03761-3. PMID 34934115
- [Background] Acil AA, Dogan S, Dogan O. The effects of physical exercises to mental state and quality of life in patients with schizophrenia. J Psychiatr Ment Health Nurs. 2008 Dec;15(10):808-15. doi: 10.1111/j.1365-2850.2008.01317.x. PMID 19012672
- [Background] Zschucke E, Gaudlitz K, Strohle A. Exercise and physical activity in mental disorders: clinical and experimental evidence. J Prev Med Public Health. 2013 Jan;46 Suppl 1(Suppl 1):S12-21. doi: 10.3961/jpmph.2013.46.S.S12. Epub 2013 Jan 30. PMID 23412549
- [Background] Gray R, Hardy S, Anderson KH. Physical health and severe mental illness: if we don't do something about it, who will? Int J Ment Health Nurs. 2009 Oct;18(5):299-300. doi: 10.1111/j.1447-0349.2009.00640.x. No abstract available. PMID 19740138
- [Background] Dimeo F, Bauer M, Varahram I, Proest G, Halter U. Benefits from aerobic exercise in patients with major depression: a pilot study. Br J Sports Med. 2001 Apr;35(2):114-7. doi: 10.1136/bjsm.35.2.114. PMID 11273973
- [Background] Curcic D, Stojmenovic T, Djukic-Dejanovic S, Dikic N, Vesic-Vukasinovic M, Radivojevic N, Andjelkovic M, Borovcanin M, Djokic G. Positive impact of prescribed physical activity on symptoms of schizophrenia: randomized clinical trial. Psychiatr Danub. 2017 Dec;29(4):459-465. doi: 10.24869/psyd.2017.459. PMID 29197203
- [Background] Ribeiro T, Fleury MJ, Granieri E, Castellazzi M, Martini F, Mazzoni E, Coursaget P, Tognon M. Investigation of the prevalence of antibodies against neurotropic polyomaviruses BK, JC and SV40 in sera from patients affected by multiple sclerosis. Neurol Sci. 2010 Aug;31(4):517-21. doi: 10.1007/s10072-010-0353-y. Epub 2010 Jun 15. PMID 20552238
- [Background] Cerini T, Hilfiker R, Riegler TF, Felsch QTM. 12 weeks high intensity interval training versus moderate intensity continuous training in chronic low back pain subjects: a randomised single-blinded feasibility study. Arch Physiother. 2022 May 2;12(1):12. doi: 10.1186/s40945-022-00136-3. PMID 35491417
- [Background] Ramos JS, Dalleck LC, Tjonna AE, Beetham KS, Coombes JS. The impact of high-intensity interval training versus moderate-intensity continuous training on vascular function: a systematic review and meta-analysis. Sports Med. 2015 May;45(5):679-92. doi: 10.1007/s40279-015-0321-z. PMID 25771785
- [Background] Wewege M, van den Berg R, Ward RE, Keech A. The effects of high-intensity interval training vs. moderate-intensity continuous training on body composition in overweight and obese adults: a systematic review and meta-analysis. Obes Rev. 2017 Jun;18(6):635-646. doi: 10.1111/obr.12532. Epub 2017 Apr 11. PMID 28401638
- [Background] Lunt H, Draper N, Marshall HC, Logan FJ, Hamlin MJ, Shearman JP, Cotter JD, Kimber NE, Blackwell G, Frampton CM. High intensity interval training in a real world setting: a randomized controlled feasibility study in overweight inactive adults, measuring change in maximal oxygen uptake. PLoS One. 2014 Jan 13;9(1):e83256. doi: 10.1371/journal.pone.0083256. eCollection 2014. PMID 24454698
- [Background] Batacan RB Jr, Duncan MJ, Dalbo VJ, Tucker PS, Fenning AS. Effects of high-intensity interval training on cardiometabolic health: a systematic review and meta-analysis of intervention studies. Br J Sports Med. 2017 Mar;51(6):494-503. doi: 10.1136/bjsports-2015-095841. Epub 2016 Oct 20. PMID 27797726
- [Background] Atan T, Karavelioglu Y. Effectiveness of High-Intensity Interval Training vs Moderate-Intensity Continuous Training in Patients With Fibromyalgia: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1865-1876. doi: 10.1016/j.apmr.2020.05.022. Epub 2020 Jun 22. PMID 32585169
- [Background] Wen D, Utesch T, Wu J, Robertson S, Liu J, Hu G, Chen H. Effects of different protocols of high intensity interval training for VO2max improvements in adults: A meta-analysis of randomised controlled trials. J Sci Med Sport. 2019 Aug;22(8):941-947. doi: 10.1016/j.jsams.2019.01.013. Epub 2019 Jan 29. PMID 30733142
- [Background] Botta RM, Palermi S, Tarantino D. High-intensity interval training for chronic pain conditions: a narrative review. J Exerc Rehabil. 2022 Feb 24;18(1):10-19. doi: 10.12965/jer.2142718.359. eCollection 2022 Feb. PMID 35356137
- [Background] Nybo L, Sundstrup E, Jakobsen MD, Mohr M, Hornstrup T, Simonsen L, Bulow J, Randers MB, Nielsen JJ, Aagaard P, Krustrup P. High-intensity training versus traditional exercise interventions for promoting health. Med Sci Sports Exerc. 2010 Oct;42(10):1951-8. doi: 10.1249/MSS.0b013e3181d99203. PMID 20195181
- [Background] Kessler HS, Sisson SB, Short KR. The potential for high-intensity interval training to reduce cardiometabolic disease risk. Sports Med. 2012 Jun 1;42(6):489-509. doi: 10.2165/11630910-000000000-00000. PMID 22587821
- [Background] Wu ZJ, Wang ZY, Gao HE, Zhou XF, Li FH. Impact of high-intensity interval training on cardiorespiratory fitness, body composition, physical fitness, and metabolic parameters in older adults: A meta-analysis of randomized controlled trials. Exp Gerontol. 2021 Jul 15;150:111345. doi: 10.1016/j.exger.2021.111345. Epub 2021 Apr 6. PMID 33836261
- [Background] Chin EC, Yu AP, Lai CW, Fong DY, Chan DK, Wong SH, Sun F, Ngai HH, Yung PSH, Siu PM. Low-Frequency HIIT Improves Body Composition and Aerobic Capacity in Overweight Men. Med Sci Sports Exerc. 2020 Jan;52(1):56-66. doi: 10.1249/MSS.0000000000002097. PMID 31343521
- [Background] Nakahara H, Ueda SY, Miyamoto T. Low-frequency severe-intensity interval training improves cardiorespiratory functions. Med Sci Sports Exerc. 2015 Apr;47(4):789-98. doi: 10.1249/MSS.0000000000000477. PMID 25137370
- [Background] Sculthorpe NF, Herbert P, Grace F. One session of high-intensity interval training (HIIT) every 5 days, improves muscle power but not static balance in lifelong sedentary ageing men: A randomized controlled trial. Medicine (Baltimore). 2017 Feb;96(6):e6040. doi: 10.1097/MD.0000000000006040. PMID 28178145
- [Background] van Baak MA, Pramono A, Battista F, Beaulieu K, Blundell JE, Busetto L, Carraca EV, Dicker D, Encantado J, Ermolao A, Farpour-Lambert N, Woodward E, Bellicha A, Oppert JM. Effect of different types of regular exercise on physical fitness in adults with overweight or obesity: Systematic review and meta-analyses. Obes Rev. 2021 Jul;22 Suppl 4(Suppl 4):e13239. doi: 10.1111/obr.13239. Epub 2021 May 3. PMID 33939229
- [Background] Martland R, Mondelli V, Gaughran F, Stubbs B. Can high-intensity interval training improve physical and mental health outcomes? A meta-review of 33 systematic reviews across the lifespan. J Sports Sci. 2020 Feb;38(4):430-469. doi: 10.1080/02640414.2019.1706829. Epub 2019 Dec 31. PMID 31889469
- [Background] Wu MH, Lee CP, Hsu SC, Chang CM, Chen CY. Effectiveness of high-intensity interval training on the mental and physical health of people with chronic schizophrenia. Neuropsychiatr Dis Treat. 2015 May 25;11:1255-63. doi: 10.2147/NDT.S81482. eCollection 2015. PMID 26060400
- [Background] Asztalos M, De Bourdeaudhuij I, Cardon G. The relationship between physical activity and mental health varies across activity intensity levels and dimensions of mental health among women and men. Public Health Nutr. 2010 Aug;13(8):1207-14. doi: 10.1017/S1368980009992825. Epub 2009 Dec 17. PMID 20018121
- [Background] Engh JA, Andersen E, Holmen TL, Martinsen EW, Mordal J, Morken G, Egeland J. Effects of high-intensity aerobic exercise on psychotic symptoms and neurocognition in outpatients with schizophrenia: study protocol for a randomized controlled trial. Trials. 2015 Dec 8;16:557. doi: 10.1186/s13063-015-1094-2. PMID 26646670
- [Background] Romain AJ, Fankam C, Karelis AD, Letendre E, Mikolajczak G, Stip E, Abdel-Baki A. Effects of high intensity interval training among overweight individuals with psychotic disorders: A randomized controlled trial. Schizophr Res. 2019 Aug;210:278-286. doi: 10.1016/j.schres.2018.12.021. Epub 2018 Dec 28. PMID 30595443
- [Background] Plag J, Schmidt-Hellinger P, Klippstein T, Mumm JLM, Wolfarth B, Petzold MB, Strohle A. Working out the worries: A randomized controlled trial of high intensity interval training in generalized anxiety disorder. J Anxiety Disord. 2020 Dec;76:102311. doi: 10.1016/j.janxdis.2020.102311. Epub 2020 Sep 24. PMID 33007710
- [Background] Andersen E, Bang-Kittilsen G, Bigseth TT, Egeland J, Holmen TL, Martinsen EW, Stensrud T, Engh JA. Effect of high-intensity interval training on cardiorespiratory fitness, physical activity and body composition in people with schizophrenia: a randomized controlled trial. BMC Psychiatry. 2020 Aug 27;20(1):425. doi: 10.1186/s12888-020-02827-2. PMID 32854688
- [Background] Gilson ND, Andersson D, Papinczak ZE, Rutherford Z, John J, Coombes JS, Brown WJ. High intensity and sprint interval training, and work-related cognitive function in adults: A systematic review. Scand J Med Sci Sports. 2023 Jun;33(6):814-833. doi: 10.1111/sms.14349. Epub 2023 Mar 20. PMID 36916717
- [Background] Bang-Kittilsen G, Engh JA, Holst R, Holmen TL, Bigseth TT, Andersen E, Mordal J, Egeland J. High-intensity interval training may reduce depressive symptoms in individuals with schizophrenia, putatively through improved VO2max: A randomized controlled trial. Front Psychiatry. 2022 Aug 4;13:921689. doi: 10.3389/fpsyt.2022.921689. eCollection 2022. PMID 36003983
- [Background] Korman N, Armour M, Chapman J, Rosenbaum S, Kisely S, Suetani S, Firth J, Siskind D. High Intensity Interval training (HIIT) for people with severe mental illness: A systematic review & meta-analysis of intervention studies- considering diverse approaches for mental and physical recovery. Psychiatry Res. 2020 Feb;284:112601. doi: 10.1016/j.psychres.2019.112601. Epub 2019 Nov 28. PMID 31883740
- [Background] Patel V, Saxena S, Lund C, Thornicroft G, Baingana F, Bolton P, Chisholm D, Collins PY, Cooper JL, Eaton J, Herrman H, Herzallah MM, Huang Y, Jordans MJD, Kleinman A, Medina-Mora ME, Morgan E, Niaz U, Omigbodun O, Prince M, Rahman A, Saraceno B, Sarkar BK, De Silva M, Singh I, Stein DJ, Sunkel C, UnUtzer J. The Lancet Commission on global mental health and sustainable development. Lancet. 2018 Oct 27;392(10157):1553-1598. doi: 10.1016/S0140-6736(18)31612-X. Epub 2018 Oct 9. No abstract available. PMID 30314863
- [Background] Henares Montiel J, Ruiz-Perez I, Sordo L. [Mental health in Spain and differences by sex, and by autonomous communities]. Gac Sanit. 2020 Mar-Apr;34(2):114-119. doi: 10.1016/j.gaceta.2019.03.002. Epub 2019 May 1. Spanish. PMID 31053452
- [Background] Wight D, Wimbush E, Jepson R, Doi L. Six steps in quality intervention development (6SQuID). J Epidemiol Community Health. 2016 May;70(5):520-5. doi: 10.1136/jech-2015-205952. Epub 2015 Nov 16. PMID 26573236
- [Background] Scherr J, Wolfarth B, Christle JW, Pressler A, Wagenpfeil S, Halle M. Associations between Borg's rating of perceived exertion and physiological measures of exercise intensity. Eur J Appl Physiol. 2013 Jan;113(1):147-55. doi: 10.1007/s00421-012-2421-x. Epub 2012 May 22. PMID 22615009
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Alos F, Colomer MA, Martin-Cantera C, Solis-Munoz M, Bort-Roig J, Saigi I, Chirveches-Perez E, Sola-Gonfaus M, Molina-Aragones JM, Puig-Ribera A. Effectiveness of a healthcare-based mobile intervention on sedentary patterns, physical activity, mental well-being and clinical and productivity outcomes in office employees with type 2 diabetes: study protocol for a randomized controlled trial. BMC Public Health. 2022 Jun 29;22(1):1269. doi: 10.1186/s12889-022-13676-x. PMID 35768818
- [Background] Zupancic V, Pahor M, Kogovsek T. Focus Group in Community Mental Health Research: Need for Adaption. Community Ment Health J. 2019 Jan;55(1):168-179. doi: 10.1007/s10597-018-0271-7. Epub 2018 Apr 27. PMID 29704087
- [Background] Vancampfort D, Firth J, Schuch FB, Rosenbaum S, Mugisha J, Hallgren M, Probst M, Ward PB, Gaughran F, De Hert M, Carvalho AF, Stubbs B. Sedentary behavior and physical activity levels in people with schizophrenia, bipolar disorder and major depressive disorder: a global systematic review and meta-analysis. World Psychiatry. 2017 Oct;16(3):308-315. doi: 10.1002/wps.20458. PMID 28941119
- [Background] Stamatakis E, Huang BH, Maher C, Thogersen-Ntoumani C, Stathi A, Dempsey PC, Johnson N, Holtermann A, Chau JY, Sherrington C, Daley AJ, Hamer M, Murphy MH, Tudor-Locke C, Gibala MJ. Untapping the Health Enhancing Potential of Vigorous Intermittent Lifestyle Physical Activity (VILPA): Rationale, Scoping Review, and a 4-Pillar Research Framework. Sports Med. 2021 Jan;51(1):1-10. doi: 10.1007/s40279-020-01368-8. PMID 33108651
- [Background] Islam H, Gibala MJ, Little JP. Exercise Snacks: A Novel Strategy to Improve Cardiometabolic Health. Exerc Sport Sci Rev. 2022 Jan 1;50(1):31-37. doi: 10.1249/JES.0000000000000275. PMID 34669625
- [Background] Stamatakis E, Ahmadi MN, Gill JMR, Thogersen-Ntoumani C, Gibala MJ, Doherty A, Hamer M. Association of wearable device-measured vigorous intermittent lifestyle physical activity with mortality. Nat Med. 2022 Dec;28(12):2521-2529. doi: 10.1038/s41591-022-02100-x. Epub 2022 Dec 8. PMID 36482104
- [Derived] Caro-Crous M, Santos JM, Jabardo-Camprubi G, Brown WJ, Puig-Ribera A. Intermittent-vigorous intensity physical activity as a strategy for recovery in severe mental illness: study protocol for a pragmatic clinical trial. BMJ Open. 2025 Dec 11;15(12):e107357. doi: 10.1136/bmjopen-2025-107357. PMID 41381109